CLINICAL TRIAL: NCT02813018
Title: The Impact of Preemptive Epidural Analgesia on Acute Postoperative Pain in Pediatric Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2016-0322
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Pediatric Surgical Patients; Preemptive Epidural Analgesia
Keywords: child; analgesia; epidural; pain; postoperative; orthopedics
MeSH Terms: conditions — Agnosia; Pain | interventions — Ropivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- preemptive group (Experimental): Group who will be received ropivacaine bolus and continous infusion 5 minutes before skin incision.
  Interventions: Procedure: 0.2 ml/kg of 0.2% ropivacaine
- saline group (Placebo Comparator): Group who will be received saline bolus and continous infusion 5 minutes before skin incision
  Interventions: Procedure: 0.2mg/kg of Normal Saline

INTERVENTIONS:
Procedure: 0.2 ml/kg of 0.2% ropivacaine — In the preemptive group, 5 minutes before skin incision, the epidural catheter is dosed with 0.2 ml/kg of 0.2% ropivacaine, followed by continuous infusion of 5 minutes before skin incision at 0.2 ml/kg/h.
  Arms: preemptive group
Procedure: 0.2mg/kg of Normal Saline — In the saline group, 5 minutes before skin incision, the epidural catheter is dosed with 0.2 ml/kg of normal saline, followed by continuous infusion of 5 minutes before skin incision at 0.2 ml/kg/h.
  Arms: saline group

SUMMARY:
Management of postoperative pain is critical in the pediatric patients, however, safe and effective analgesia for pediatric surgical patients remains a challenge. Preemptive analgesia is based on preventing a prolonged change in central nervous system function by blocking afferent input before the surgical stimulation may evoke central sensitization and aggravate amplification and prolongation of postoperative pain. However, the clinical efficacy of preemptive analgesia is still controversial. In this study, the investigators aim to assess the impact of preemptive epidural analgesia on postoperative pain in pediatric patients for corrective osteotomy of the lower extremities expecting severe postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (3-12 years of age) scheduled for corrective osteotomy of the lower extremities
* ASA class I and II

Exclusion Criteria:

* Coagulopathy
* Neurological disease
* Allergy to local anesthetics or contraindication to use of ropivacaine
* Infection at the site of epidural catheter insertion

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
FLACC scale score (Face, Legs, Activity, Cry, Consolability) | 0-6 hours after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025